CLINICAL TRIAL: NCT06966206
Title: Multiprofen-CC to Reduce Pain in Hand Arthritis (MRP-HAND): A Crossover Randomized Controlled Trial
Brief Title: Multiprofen-CC to Reduce Pain in Hand Arthritis
Acronym: MRP-HAND
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Research Institute of St Joe's Hamilton (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRP-HAND
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-04

CONDITIONS: Hand Osteoarthritis
Keywords: hand osteoarthritis; osteoarthritis; arthritis; topical; multiprofen
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Intervention Model Description: 2x2 crossover randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiprofen-CC™ (Experimental): Multiprofen-CC™ [ketoprofen (10%), baclofen (5%), amitriptyline (2%), and lidocaine (5%)] Dose: 1.0g, 3 times per day for 2 weeks
  Interventions: Drug: Multiprofen-CC™ plus standard treatment
- Placebo (Placebo Comparator): The placebo is the base cream with no medicinal ingredients Dose: 1.0g, 3 times per day for 2 weeks
  Interventions: Other: Placebo plus standard treatment

INTERVENTIONS:
Drug: Multiprofen-CC™ plus standard treatment — Standard care pain medications and topical Multiprofen-CC™ (1g TID) for 2 weeks
  Arms: Multiprofen-CC™
Other: Placebo plus standard treatment — Standard care pain medications and visually identical topical placebo (1g TID) for 2 weeks
  Arms: Placebo

SUMMARY:
This clinical trial aims to find out if using 1 gram of Multiprofen-CC cream on the hands three times a day for 4 weeks can help reduce pain in adults with hand osteoarthritis, compared to a placebo (a cream with no active medicine). The research team will also look at how Multiprofen-CC affects hand function, opioid use, and how patients feel about their overall improvement. In addition, the research team will keep track of any side effects.

Participants will:

* Use both Multiprofen-CC and a placebo (a cream with no active medicine) during the study, in a random order.
* Be asked to apply 1 gram of cream to their hands three times a day for 2 weeks, following the manufacturer's instructions.
* Attend a visit before starting the study, after 2 weeks, and after 6 weeks.
* Report any symptoms they experience during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+)
* Have been diagnosed with hand osteoarthritis according to American College of Rheumatology criteria
* Experience pain and/or loss of function in one or both hands that interferes with daily life
* Provide informed consent

Exclusion Criteria:

* Unable to consent
* Unable or unwilling to follow study protocol
* Known allergy or contraindication to any of the study drugs or their ingredients
* Have open wounds/cuts and/or skin conditions on the hand area
* Pregnant or breastfeeding
* History of impaired kidney or liver function
* Rheumatoid or other inflammatory arthropathy
* Hand surgery within the past 6 months or planned within the study period.
* Use daily opioids (other than short acting codeine) for a chronic pain condition other than hand arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | baseline [week 0] and weeks 2, 4, and 6
  Average pain intensity will be measured using a 0-10 Numeric Rating Scale (NRS), where 0 represents "no pain" and 10 represents "worst imaginable pain." Scores are collected before and after each treatment period. Higher scores indicate greater pain intensity and thus a worse outcome.

SECONDARY OUTCOMES:
Pain interference | weeks 2, 4 and 6
  Measured using the 7 pain interference items from the Brief Pain Inventory - Short Form (BPI-SF). Each item is rated on a scale from 0 to 10, where 0 indicates "does not interfere" and 10 indicates "completely interferes." The total pain interference score is calculated as the average of the seven items, with a minimum possible value of 0 and a maximum of 10. Higher scores indicate worse pain interference and thus a worse outcome.
Hand function | weeks 2, 4 and 6
  Measured using the Michigan Hand Outcomes Questionnaire (MHQ), a validated instrument assessing hand function, activities of daily living, work performance, pain, aesthetics, and patient satisfaction. The total score ranges from 0 to 100, with higher scores representing better overall hand function and patient-reported outcomes.
Patients reported improvement | weeks 2, 4 and 6
  Measured using the Patient Global Impression of Change (PGIC) scale, a single-item, patient-reported measure of overall improvement. The scale ranges from 1 to 7, where 1 indicates "very much improved" and 7 indicates "very much worse." Lower scores represent better outcomes.
Safety - adverse events | through study completion, an average of 6 weeks
  Hand-related and medication-related serious and non-serious adverse events

OTHER OUTCOMES:
Thumb Disability (exploratory outcome) | weeks 2, 4, and 6
  Patients with thumb carpometacarpal (CMC) osteoarthritis will complete the Thumb Disability Examination (TDX), a patient-reported outcome measure that assesses functional disability related to thumb CMC osteoarthritis. Scores range from 0 to 100, with higher scores indicating greater disability and therefore a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Levis, MD, MSc, FRCS(C), Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No